CLINICAL TRIAL: NCT05468918
Title: Real World Perspectives on Advancements in Hearing Aid Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-2855
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded as to which device they were wearing during the lab testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Participants tested with comparator devices first, then Audeo Lumity devices (Experimental): All participants who completed speech in noise testing in the lab with the comparator devices first, and then the Audeo Lumity devices.
  Interventions: Device: Phonak Audeo previous generation hearing aids; Device: Phonak Audeo Lumity hearing aids
- Participants who were tested with Audeo Lumity first, then comparator devices (Experimental): All participants who completed speech in noise testing in the lab with the Audeo Lumity devices first, and then the comparator devices.
  Interventions: Device: Phonak Audeo previous generation hearing aids; Device: Phonak Audeo Lumity hearing aids

INTERVENTIONS:
Device: Phonak Audeo previous generation hearing aids — Receiver-in-canal (RIC) hearing aids with universal earpieces
Device: Phonak Audeo Lumity hearing aids — Receiver-in-canal (RIC) hearing aids with universal earpieces

SUMMARY:
This study will compare different microphone technologies in a noisy environment when the dominant speaker is at the front, back, left, or right side of the listener.

DETAILED DESCRIPTION:
Understanding speech in a noisy environment can be difficult for people with hearing loss even with hearing aids. Hearing aid manufacturers have implanted various methods (i.e., directional micro-phones, noise reduction, noise cancelers) to try to improve the signal-to-noise ratio (SNR) to increase the speech understanding in these difficult listening situations.

This study is evaluating different microphone technologies to determine listening effort when speech is to the back or side of the listener in noisy environment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate sensorineural hearing loss
* Experienced hearing aid user
* Has a significant other/communication partner that can fill out a questionnaire about hearing aid performance during the home trial
* Smartphone user for receiving study alerts

Exclusion Criteria:

* Cognitive impairment
* Not willing to wear hearing aid

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Tested With Comparator Devices First, Than Audeo Lumity Devices: All participants who completed speech in noise testing in the lab with the comparator devices first, and then the Audeo Lumity devices.
  Phonak Audeo previous generation hearing aids: Receiver-in-canal (RIC) hearing aids with universal earpieces Phonak Audeo Lumity hearing aids: Receiver-in-canal (RIC) hearing aids with universal earpieces
- Participants Tested With Audeo Lumity First, Than Comparator Devices: All participants who completed speech in noise testing in the lab with the Audeo Lumity devices first, and then the comparator devices.
  Phonak Audeo previous generation hearing aids: Receiver-in-canal (RIC) hearing aids with universal earpieces Phonak Audeo Lumity hearing aids: Receiver-in-canal (RIC) hearing aids with universal earpieces
Period: Overall Study
Arm/Group | Participants Tested With Comparator Devices First, Than Audeo Lumity Devices | Participants Tested With Audeo Lumity First, Than Comparator Devices
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Tested With Both Devices.: Participants who complete lab testing and home trials with both the comparator devices and the Audeo Lumity devices.
Arm/Group | All Participants Tested With Both Devices.
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 75 [65 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Speech in Noise Test
Description: A speech in noise test in which participants repeat words which are presented in the presence of background noise. In a 12-speaker array, speech is presented from speakers either on the left side of the participant (-90 degrees) or from behind the participant (180 degrees) while background noise is presented from remaining speakers. Scores are calculated as the number of words correctly repeated and expressed as a percentage. A higher percentage or score is better.
Time Frame: Day 1 of study
Measure: Mean (Full Range); unit: percentage of correct responses
Arm/Group | All Participants Tested With Both Devices.
Number analyzed (Participants) | 14
percentage of correct responses
  Percent correct with Lumity devices | 84.84 [52.5 to 99]
  Percent correct with comparator devices | 77.16 [24 to 98.5]
Statistical Analysis 1: Comparison: All Participants Tested With Both Devices; Test type: Other; p = 0.002, ANOVA

2. Primary Outcome: Subjective Perception of Listening Effort
Description: Following the speech in noise testing in the lab, participants rated their listening effort on a scale from 1 to 10, with 1 = no effort and 10 = a lot of effort. In this case, a lower rating is better as it indicates less perceived listening effort.
Time Frame: Day 1 of study
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | All Participants Tested With Both Devices.
Number analyzed (Participants) | 14
score on a scale
  Listening effort rating with Lumity devices | 5.82 [1 to 10]
  Listening effort rating with comparator devices | 6.82 [3 to 10]
Statistical Analysis 1: Comparison: All Participants Tested With Both Devices; Test type: Other; p = 0.023, ANOVA

ADVERSE EVENTS:
Time Frame: 4 Weeks. Participants had one day testing in the lab followed by a two week home trial.
Groups:
- All Participants Who Wore Comparator Devices: All participants who completed lab testing and home trial with the Comparator devices.
  Phonak Audeo previous generation hearing aids: Receiver-in-canal (RIC) hearing aids with universal earpieces
- All Participants Who Wore Audeo Lumity Devices: All participants who completed lab testing and home trial with the Audeo Lumity devices.
  Phonak Audeo Lumity hearing aids: Receiver-in-canal (RIC) hearing aids with universal earpieces
Arm/Group | All Participants Who Wore Comparator Devices | All Participants Who Wore Audeo Lumity Devices
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05468918/Prot_SAP_000.pdf